CLINICAL TRIAL: NCT04631172
Title: Evaluation of Covid-19 Anxiety and Phobia Levels of the Parents of Pediatric Patients
Brief Title: Covid-19 Anxiety and Phobia Levels of the Parents
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Faruk Cicekci, Principal investigator, Selcuk University
Other Study IDs: farukcicekci
Record Dates: First submitted 2020-11-14; First posted 2020-11-17 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: SARS-CoV-2; Anxiety and Fear; Parents
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Coronavirus Anxiety Scale , COVID-19 Phobia Scale — Using two questionnaire completed in face-to-face interviews Participants were asked the Coronavirus Anxiety Scale (CAS), and the COVID-19 Phobia Scale (C19P-S).

SUMMARY:
A pandemic that originated in the Wuhan region of China in December 2019 was detected as a new type of coronavirus disease called coronavirus 2019 (COVID-19). In the first phase of the outbreak, specialists explained ways to maintain physical health . However, pediatric surgical procedures and anesthesia applications continued during this period. Surgery in pediatric patients is an unpleasant and potentially 'threatening' experience, often followed by preoperative anxiety due to the child's illness, hospitalization, fear of anesthesia - especially the time of anesthesia induction - and the surgery itself . Anesthesia is a stressful procedure for the child and the entire family. Both the COVID-19 pandemic and the surgical procedure are reflected in the symptoms of anxiety, fear or acute stress disorder for children and their families. As the disease spread, investigators started to emphasize the importance of protecting mental health. Identifying factors that contribute to significant preoperative anxiety levels in pediatric patients and their parents can help healthcare professionals choose the most appropriate from a variety of alternative strategies for anxiety control. This study was planned to evaluate the COVID-19 anxiety and phobia levels of the parents of pediatric patients are scheduled to undergo surgery under general anesthesia in Turkey.

DETAILED DESCRIPTION:
The population of the study was created from the parents of pediatric patients who were scheduled for surgery under general anesthesia between May 2020 and September 2020 at Selcuk University Department of Anesthesiology and Reanimation. The data were obtained through face-to-face interviews before the child was taken to surgery after the necessary explanations were made to the parents of the children by the researchers. To enable the parents to answer the questions easily, a separate room in the relevant clinic was used for the interviews. The characteristics of the children and parents, supplementary data of the parents regarding the child's illness, and contact information were obtained. Participants were asked to complete a sociodemographic data form, the Coronavirus Anxiety Scale (CAS), and the COVID-19 Phobia Scale (C19P-S).

ELIGIBILITY:
Inclusion Criteria:

* Parents of pediatric patients with American Society of Anesthesiologists classification (ASA) I-II, aged 1-12 years who were administered anesthesia to undergo surgery were included in the study.

Exclusion Criteria:

* Parents of children with ASA III or higher risk, expected to have difficult intubation, serious complications related to intraoperative surgery or anesthesia (e.g. respiratory depression, myocardial depression, cardiac arrhythmia, bronchospasm, laryngospasm, anaphylactic reaction, hypotension, bleeding), and could not communicate were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The parents of pediatric patients who were scheduled to undergo surgery under general anesthesia in Turkey
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Coronavirus Anxiety Scale (CAS) | 5 months
  The Coronavirus Anxiety Scale (CAS), which was developed by Lee and validated in Turkish by Evren et al., was used to evaluate the COVID-19 anxiety level. In the validation study, the Cronbach's alpha of the Turkish version of CAS was 0.87. This results of the study showed that the CAS was highly reliable. CAS is a 5-point Likert-type scale. The scale consists of five questions and one dimension. Scoring of the scale is evaluated as 0 = never, 1 = rare, less than a day or two, 2 = a few days, 3 = more than a week, and 4 = almost every day in the last two weeks. The total score ranges from 0 to 20. Lee determined the CAS cut-off score of 9 to distinguish those with dysfunctional anxiety from those without anxiety.
COVID 19 phobia scale (C19P-S) | 5 months
  COVID 19 phobia scale (C19P-S) is a 20-item, 4-subdimension (psychological, somatic, social and economic) scale in which items are answered in a 5-point response format developed by Arpacı et al. 7 to measure the phobia that may develop against COVID-19. In the validation study, the Cronbach's alpha of the Turkish version of C19P-S was 0.92. In the present study, Cronbach's alpha was 0.94. The results of the study demonstrated that the C19P-S was exceptionally reliable. The scale items are rated between 1 "strongly disagree" and 5, "strongly agree. Sub-dimension scores are obtained by the sum of the points of the answers given to the items belonging to that sub-dimension, while the total C19P-S score is obtained by the total of the subdimension scores, ranging between 20 and 100 points.

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Cicekci, Principal Investigator — Selcuk University, School of Medicine, Department of Anesthesiology and Intensive Care
Locations (1):
- Selcuk University, School of Medicine, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided